CLINICAL TRIAL: NCT03348930
Title: Tolcapone Treatment of Obsessive Compulsive Disorder: A Double-Blind, Placebo-Controlled, Cross-Over Pilot Study
Brief Title: Tolcapone in Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-1379
Record Dates: First submitted 2017-11-15; First posted 2017-11-21 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tolcapone (Experimental): Each subject will have a 4 week treatment phase with Tolcapone
  Interventions: Drug: Tolcapone 200 MG
- Placebo (Placebo Comparator): 4 week placebo phase before or after Tolcapone phase depending on randomization.
  Interventions: Drug: Tolcapone 200 MG

INTERVENTIONS:
Drug: Tolcapone 200 MG — All eligible study subjects will go through a 2-week treatment phase during which they will begin tolcapone at 100mg twice a day.
  Other Names: No other names

SUMMARY:
The proposed study will consist of a 5-week double-blind cross-over study trial of tolcapone in 20 people (ages 18-65). The study will be divided into an initial 2 week phase and a second 2 week phase, with one of the 2 week phases consisting of active treatment with tolcapone, and the other 2 week phase consisting of inactive placebo treatment. There will be a one-week wash-out phase between the 2-week treatment phases. Participants will be randomized to receive either tolcapone or placebo during the first 2 week phase on a 1:1 basis. This blinding will be maintained by the IDS pharmacy at the University of Chicago.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy and safety of tolcapone in adults with obsessive compulsive disorder (OCD). The hypothesis to be tested is that tolcapone will be more effective and well tolerated in adults with OCD compared to placebo. The proposed study will provide needed data on the treatment of a disabling disorder where current treatments are often ineffective.

The primary aim of this application is to conduct a randomized placebo-controlled pharmacotherapy trial using tolcapone in 20 participants with OCD. The study will consist of two phases: a 2 week active treatment phase with tolcapone, a one-week wash-out phase, and a 2 week placebo phase. The subjects will be randomized to either receive tolcapone or placebo treatment in the first 2 weeks, and the other during the remaining 2 week phase.

This will be one of few studies assessing the use of pharmacotherapy for the treatment of OCD in adults. Assessing the efficacy and safety of tolcapone will help inform clinicians about additional treatment options for adults suffering from this disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18-65;
2. Diagnosis of current OCD based on DSM-5 criteria and confirmed using the clinician-administered Structured Clinical Interview for DSM-5 (SCID);
3. Able and willing to provide written consent for participation.

Exclusion Criteria:

1. Unstable medical illness, including liver disease, as determined by the investigator;
2. History of seizures;
3. Clinically significant suicidality (defined by the Columbia Suicide Severity Rating Scale);
4. Baseline score of ≥17 on the Hamilton Depression Rating Scale (17-item HDRS);
5. Lifetime history of bipolar disorder type I or II, schizophrenia, autism, any psychotic disorder, or any substance use disorder;
6. Initiation of psychotherapy or behavior therapy within 3 months prior to study baseline;
7. Previous treatment with tolcapone;
8. Any history of psychiatric hospitalization in the past year;
9. Currently pregnant (confirmed by urine pregnancy test)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD,MD,MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saxena S, Rauch SL. Functional neuroimaging and the neuroanatomy of obsessive-compulsive disorder. Psychiatr Clin North Am. 2000 Sep;23(3):563-86. doi: 10.1016/s0193-953x(05)70181-7. PMID 10986728
- [Background] Baxter LR Jr, Phelps ME, Mazziotta JC, Guze BH, Schwartz JM, Selin CE. Local cerebral glucose metabolic rates in obsessive-compulsive disorder. A comparison with rates in unipolar depression and in normal controls. Arch Gen Psychiatry. 1987 Mar;44(3):211-8. doi: 10.1001/archpsyc.1987.01800150017003. PMID 3493749
- [Background] Milad MR, Rauch SL. Obsessive-compulsive disorder: beyond segregated cortico-striatal pathways. Trends Cogn Sci. 2012 Jan;16(1):43-51. doi: 10.1016/j.tics.2011.11.003. Epub 2011 Dec 2. PMID 22138231
- [Background] Graybiel AM, Rauch SL. Toward a neurobiology of obsessive-compulsive disorder. Neuron. 2000 Nov;28(2):343-7. doi: 10.1016/s0896-6273(00)00113-6. No abstract available. PMID 11144344
- [Background] Piras F, Piras F, Caltagirone C, Spalletta G. Brain circuitries of obsessive compulsive disorder: a systematic review and meta-analysis of diffusion tensor imaging studies. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2856-77. doi: 10.1016/j.neubiorev.2013.10.008. Epub 2013 Oct 28. PMID 24177038
- [Background] Menzies L, Achard S, Chamberlain SR, Fineberg N, Chen CH, del Campo N, Sahakian BJ, Robbins TW, Bullmore E. Neurocognitive endophenotypes of obsessive-compulsive disorder. Brain. 2007 Dec;130(Pt 12):3223-36. doi: 10.1093/brain/awm205. Epub 2007 Sep 13. PMID 17855376
- [Background] Chamberlain SR, Menzies L, Hampshire A, Suckling J, Fineberg NA, del Campo N, Aitken M, Craig K, Owen AM, Bullmore ET, Robbins TW, Sahakian BJ. Orbitofrontal dysfunction in patients with obsessive-compulsive disorder and their unaffected relatives. Science. 2008 Jul 18;321(5887):421-2. doi: 10.1126/science.1154433. PMID 18635808
- [Background] Skoog G, Skoog I. A 40-year follow-up of patients with obsessive-compulsive disorder [see commetns]. Arch Gen Psychiatry. 1999 Feb;56(2):121-7. doi: 10.1001/archpsyc.56.2.121. PMID 10025435
- [Background] Mancebo MC, Eisen JL, Pinto A, Greenberg BD, Dyck IR, Rasmussen SA. The brown longitudinal obsessive compulsive study: treatments received and patient impressions of improvement. J Clin Psychiatry. 2006 Nov;67(11):1713-20. doi: 10.4088/jcp.v67n1107. PMID 17196050
- [Background] Blanco C, Olfson M, Stein DJ, Simpson HB, Gameroff MJ, Narrow WH. Treatment of obsessive-compulsive disorder by U.S. psychiatrists. J Clin Psychiatry. 2006 Jun;67(6):946-51. doi: 10.4088/jcp.v67n0611. PMID 16848654
- [Background] Grant JE. Clinical practice: Obsessive-compulsive disorder. N Engl J Med. 2014 Aug 14;371(7):646-53. doi: 10.1056/NEJMcp1402176. PMID 25119610
- [Background] Tunbridge EM, Bannerman DM, Sharp T, Harrison PJ. Catechol-o-methyltransferase inhibition improves set-shifting performance and elevates stimulated dopamine release in the rat prefrontal cortex. J Neurosci. 2004 Jun 9;24(23):5331-5. doi: 10.1523/JNEUROSCI.1124-04.2004. PMID 15190105
- [Background] Mier D, Kirsch P, Meyer-Lindenberg A. Neural substrates of pleiotropic action of genetic variation in COMT: a meta-analysis. Mol Psychiatry. 2010 Sep;15(9):918-27. doi: 10.1038/mp.2009.36. Epub 2009 May 5. PMID 19417742
- [Background] Apud JA, Mattay V, Chen J, Kolachana BS, Callicott JH, Rasetti R, Alce G, Iudicello JE, Akbar N, Egan MF, Goldberg TE, Weinberger DR. Tolcapone improves cognition and cortical information processing in normal human subjects. Neuropsychopharmacology. 2007 May;32(5):1011-20. doi: 10.1038/sj.npp.1301227. Epub 2006 Oct 25. PMID 17063156
- [Background] Servan-Schreiber D, Printz H, Cohen JD. A network model of catecholamine effects: gain, signal-to-noise ratio, and behavior. Science. 1990 Aug 24;249(4971):892-5. doi: 10.1126/science.2392679.
- [Background] Seamans JK, Yang CR. The principal features and mechanisms of dopamine modulation in the prefrontal cortex. Prog Neurobiol. 2004 Sep;74(1):1-58. doi: 10.1016/j.pneurobio.2004.05.006. PMID 15381316
- [Background] Malhotra AK, Kestler LJ, Mazzanti C, Bates JA, Goldberg T, Goldman D. A functional polymorphism in the COMT gene and performance on a test of prefrontal cognition. Am J Psychiatry. 2002 Apr;159(4):652-4. doi: 10.1176/appi.ajp.159.4.652. PMID 11925305
- [Background] Roussos P, Giakoumaki SG, Pavlakis S, Bitsios P. Planning, decision-making and the COMT rs4818 polymorphism in healthy males. Neuropsychologia. 2008 Jan 31;46(2):757-63. doi: 10.1016/j.neuropsychologia.2007.10.009. Epub 2007 Oct 22. PMID 18037454
- [Background] Bitsios P, Roussos P. Tolcapone, COMT polymorphisms and pharmacogenomic treatment of schizophrenia. Pharmacogenomics. 2011 Apr;12(4):559-66. doi: 10.2217/pgs.10.206. PMID 21521027
- [Background] Roussos P, Giakoumaki SG, Bitsios P. Tolcapone effects on gating, working memory, and mood interact with the synonymous catechol-O-methyltransferase rs4818c/g polymorphism. Biol Psychiatry. 2009 Dec 1;66(11):997-1004. doi: 10.1016/j.biopsych.2009.07.008. Epub 2009 Aug 22. PMID 19699472
- [Background] Forsberg M, Lehtonen M, Heikkinen M, Savolainen J, Jarvinen T, Mannisto PT. Pharmacokinetics and pharmacodynamics of entacapone and tolcapone after acute and repeated administration: a comparative study in the rat. J Pharmacol Exp Ther. 2003 Feb;304(2):498-506. doi: 10.1124/jpet.102.042846. PMID 12538800
- [Background] Blum K, Chen TJ, Meshkin B, Waite RL, Downs BW, Blum SH, Mengucci JF, Arcuri V, Braverman ER, Palomo T. Manipulation of catechol-O-methyl-transferase (COMT) activity to influence the attenuation of substance seeking behavior, a subtype of Reward Deficiency Syndrome (RDS), is dependent upon gene polymorphisms: a hypothesis. Med Hypotheses. 2007;69(5):1054-60. doi: 10.1016/j.mehy.2006.12.062. Epub 2007 Apr 30. PMID 17467918
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] Olanow CW, Watkins PB. Tolcapone: an efficacy and safety review (2007). Clin Neuropharmacol. 2007 Sep-Oct;30(5):287-94. doi: 10.1097/wnf.0b013e318038d2b6. PMID 17909307
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Sheehan DV. (1983). The Anxiety Disease. New York: Scribner's.
- [Background] Guy W (1976). ECDEU Assessment Manual for Psychopharmacology. US Dept Health, Education and Welfare publication (ADM) 76-338. Rockville, MD: National Institute of Mental Health, 218-222.

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolcapone, Then Placebo: Each subject will have a 2 week active treatment phase first with Tolcapone (100mg, twice a day), followed by a one-week washout period, followed by a 2 week treatment phase with a Tolcapone-matched placebo tablet.
- Placebo, Then Tolcapone: Each subject will have a 2 week active treatment phase first with a Tolcapone-matched placebo, followed by a one-week washout period, followed by a 2 week active treatment phase with Tolcapone (100mg, twice a day).
Period: First Intervention (2 Weeks)
Arm/Group | Tolcapone, Then Placebo | Placebo, Then Tolcapone
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Tolcapone, Then Placebo | Placebo, Then Tolcapone
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Second Intervention (2 Weeks)
Arm/Group | Tolcapone, Then Placebo | Placebo, Then Tolcapone
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tolcapone/Placebo: Each subject will have a 4 week treatment phase with Tolcapone and a 4 week placebo phase before or after Tolcapone phase depending on randomization.
  Tolcapone 200 MG: All eligible study subjects will go through a 2-week treatment phase during which they will begin tolcapone at 100mg twice a day.
Arm/Group | Tolcapone/Placebo
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12
  African American | 4
  Latino/Hispanic | 1
  Other | 2
  Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
Any psychiatric comorbidity [Count of Participants; unit: Participants]
  Yes | 9
  No | 11

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale (Y-BOCS)
Description: The entire study for the subject will last 5 weeks. Every 2 weeks and after the one week washout period the subject will take the YBOCS. The change in scores from baseline to after 5 weeks will be assessed. The scale itself assesses severity of OCD symptoms. The YBOCS scale ranges from 0 to 40, with 0 being no symptoms and 40 being severe.
Time Frame: 2 weeks (start of study to washout period OR two weeks following washout period)
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: mean change in YBOCS score
Groups:
- Tolcapone: Tolcapone 200 MG: All eligible study subjects will go through a 2-week treatment phase (either during the first two weeks or last two weeks of the study) during which they will begin tolcapone at 100mg twice a day.
- Placebo: All eligible study subjects will go through a 2-week phase (either during the first two weeks or last two weeks of the study) during which they will begin the tolcapone-matched placebo twice a day.
Arm/Group | Tolcapone | Placebo
Number analyzed (Participants) | 19 | 19
mean change in YBOCS score | -4.24 (6.20) | -1.10 (4.71)

2. Secondary Outcome: Clinical Global Impression- Severity and Improvement (CGI)
Description: The entire study for the subject will last 5 weeks. Every two weeks and after the one week washout period the subject will complete the CGI. The change in scores from baseline to after 5 weeks will be assessed. The scale itself assesses overall disorder severity on a scale from 1 to 7 with 1 being "not at all" and 7 being "among the most severe cases"
Time Frame: 2 weeks (start of study to washout period OR two weeks following washout period)
Population: Participants who fully completed Visits 2 and 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tolcapone | Placebo
Number analyzed (Participants) | 17 | 19
score on a scale | 3.78 (1.43) | 3.5 (0.90)

3. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The entire study for the subject will last 5 weeks. Every two weeks and after the one week washout period the subject will complete the SDS. The change in scores from baseline to after 5 weeks will be assessed. The scale itself assesses the level of disability from obsessive compulsive disorder (or target disorder). The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. Work/school scores range from 0 to 10, Social life scores range from 0 to 10, Family life/home responsibilities scores range from 0 to 10). Total scores are calculated by adding the scores for work/school, social life, and family life. Total scores range from a minimum of 0 to a maximum of 30 (0 unimpaired, 30 highly impaired).
Time Frame: 2 weeks (start of study to washout period OR two weeks following washout period)
Population: Subjects who completed all five weeks of the study except for one subjects who's SDS data was missing at all time points (no data to carry forward).
Measure: Mean (Standard Deviation); unit: mean change in SDS score
Arm/Group | Tolcapone | Placebo
Number analyzed (Participants) | 18 | 18
mean change in SDS score | -2.68 (4.41) | -1.97 (6.62)

4. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: Every study visit, the subject will complete the HAM-A. The change in scores from baseline to after 5 weeks will be assessed. The scale itself assesses level of anxiety. Higher scores indicate higher levels of anxiety, with 0 being no symptoms of anxiety and 30 being severe anxiety.
Time Frame: 2 weeks (start of study to washout period OR two weeks following washout period)
Population: Adults with OCD who completed the study.
Measure: Mean (Standard Deviation); unit: mean change in HAM-A score
Arm/Group | Tolcapone | Placebo
Number analyzed (Participants) | 19 | 19
mean change in HAM-A score | -1.90 (4.39) | -1.60 (4.07)

5. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: The entire study for the subject will last 5 weeks. The HAM-D will be administered at every study visit. The change in scores from baseline to after the end of the 2-week active treatment period will be assessed and the change in scores from baseline to the end of the 2-week placebo period. The scale itself assesses level of depression. The minimum score is 0 and indicates no depressive symptoms, while the highest possible score is 50. Higher total scores indicate high levels of depression. Higher scores indicate a worse outcome. Higher total scored (14-50) indicate higher levels of depression, while a score between 0-7 is considered normal.
Time Frame: 2 weeks (start of study to washout period OR two weeks following washout period)
Population: Adults with OCD who completed the 5-week study.
Measure: Mean (Standard Deviation); unit: mean change in HAM-D score
Arm/Group | Tolcapone | Placebo
Number analyzed (Participants) | 19 | 19
mean change in HAM-D score | -1.65 (3.67) | -2.00 (4.42)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, as necessary over the period of 5 week (the length of the trial).
Groups:
- Tolcapone: Subjects received 100mg of tolcapone twice a day for two weeks either starting after the baseline visit, or starting after the 1-week washout period.
- Placebo: Subjects received tolcapone-matched placebo twice a day for two weeks either starting after the baseline visit, or starting after the 1-week washout period.
Arm/Group | Tolcapone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolcapone (N=20) | Placebo (N=20)
Mild Headache (General disorders) | 1 | 0
Increased frequency in bowel movements (Gastrointestinal disorders) | 1 | 0
Blood in stool (Gastrointestinal disorders) | 1 | 0 — This was followed up and found to be haemorrhoids
Less frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Muscle aching (General disorders) | 0 | 1
Joint stiffness (General disorders) | 0 | 1
Sleep problems (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT03348930/Prot_SAP_001.pdf